CLINICAL TRIAL: NCT01992224
Title: Effect of Early Mechanical Ventilation to Severe Acute Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Erzhen Chen, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAP bundle -- MV; 12411950500 (Other Grant/Funding Number: Science and Technology Commission of Shanghai Municipality)
Record Dates: First submitted 2013-11-06; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Acute Pancreatitis; Complication of Ventilation Therapy
Keywords: severe acute pancreatitis; mechanical ventilation
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- early mechanical ventilation (Experimental): Fulfillment of three or more criteria below:
  respiratory rate > 28 per minute serum lactate > 3 mmol/L PaO2/FiO2 Index <300 mmHg SvO2 < 65% lung infiltration or atelectasis, pleural exudation
  Abbreivation: PaO2, arterial partial pressure of oxygen; FiO2, fraction of inspired oxygen; SvO2, venous oxygen saturation
  Interventions: Other: early mechanical Ventilation
- conventional mechanical ventilation (Experimental): other group who don't start early mechanical ventilation and fulfillment four criteria below: respiratory rate > 28 bpm dyspnea PaO2/FiO2 Index <200 mmHg Chest X-ray: lung infiltration exclude chronic heart failure and pulmonary disease
  Interventions: Other: Conventional Mechanical Ventilation

INTERVENTIONS:
Other: early mechanical Ventilation — Fulfillment of three or more criteria below:
  respiratory rate > 28 per minute serum lactate > 3 mmol/L PaO2/FiO2 Index <300 mmHg SvO2 < 65% lung infiltration or atelectasis, pleural exudation
  Arms: early mechanical ventilation
Other: Conventional Mechanical Ventilation — other group who don't start early mechanical ventilation and fulfillment four criteria below: respiratory rate > 28 bpm dyspnea PaO2/FiO2 Index <200 mmHg Chest X-ray: lung infiltration exclude chronic heart failure and pulmonary disease
  Arms: conventional mechanical ventilation

SUMMARY:
Acute lung injury (ALI) and acute respiratory distress syndrome(ARDS) represent the most common and earliest organ dysfunction in acute pancreatitis, presenting as dyspnea and intractable hypoxemia, with secondary bilateral pulmonary infiltrates on radiograph. And mechanical ventilation (MV) is the essential intervention to improve oxygenation. When to initiate MV remains uncertain. In this study, we aim to compare the effect of early MV and conventional MV, and we hypothesize that early MV may be a better treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pancreatitis:typical pain, increase in serum lipase or amylase, onset of abdominal pain within 72h before admission
* The diagnosis criteria of Severe Acute Pancreatitis is according to Atlanta criteria revisited in 2012
* the diagnosis of ARDS meets the criteria of Berlin definition

Exclusion Criteria:

* chronic respiratory disease as chronic obstructive pulmonary disease (COPD), asthma
* organic cardiopathy
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Mechanical Ventilation Time | 28 days

SECONDARY OUTCOMES:
the incidence of ventilation associated pneumonia | 28 days

OTHER OUTCOMES:
mortality | 60 days
the incidence other complications of mechanical ventilation | participants will be followed for the duration of hospital stay, an expected average of 2 months
  patient-mechanic desynchronization, pneumothorax, atelectasis
hospital stay | the participants will be followed till the discharge, an expected average of 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of EICU, Ruijin Hospital, Shanghai, China